CLINICAL TRIAL: NCT03940885
Title: Erector Spinae Plane Block: An Analgesic Technique as an Alternative to Transversus Abdominis Plane Block in Abdominoplasty Surgery
Brief Title: Erector Spinae Plane Block Versus Transversus Abdominis Plane Block in Abdominoplasty Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MD.19.03.155
Record Dates: First submitted 2019-05-06; First posted 2019-05-07 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Abdominoplasty
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: single-blind study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Erector spinea plane block group (Active Comparator): this group is planned for ultrasound-guided Transversus abdominis plane block
  Interventions: Procedure: Erector spinea plane block group
- Transversus abdominis plane block (Active Comparator): this group is planned for ultrasound-guided Transversus abdominis plane block
  Interventions: Procedure: Transversus abdominis plane block
- Control group (Placebo Comparator): standard general anesthesia
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Erector spinea plane block group — Which will receive ultrasound-guided erector spinea plane block bilaterally and the local anesthetic injected will be total volume 25 ml on each side consisting of 15ml of 0.5% plus 5 ml 2% lidocaine HCL plus 5 ml saline
  Arms: Erector spinea plane block group
Procedure: Transversus abdominis plane block — Which will receive ultrasound-guided Transversus Abdominis plane block bilaterally and the local anesthetic used will be total volume 25 ml on each side consisting of 15ml of 0.5% plus 5 ml 2% lidocaine HCL plus 5 ml saline
  Arms: Transversus abdominis plane block
Procedure: Control group — this group will receive only standard general anesthesia
  Arms: Control group

SUMMARY:
Abdominoplasty is one of the most popular body-contouring procedures. Patients that undergo body-contouring abdominoplasty usually have important analgesic requirements. Given the substantial incision and soft-tissue undermining associated with this procedure, postoperative pain is a concern for patients and surgeons. Previous studies have typically incorporated multiple nerve blocks to improve analgesia after abdominoplasty. Different anesthetic techniques have been developed to overcome this problem such as Epidural anesthesia, Transversus abdominis plane block either open technique or ultrasound-guided, Paravertebral block and Erector Spinea plane block. Improving postoperative pain control in this kind of surgery leads to earlier mobilization, shortened hospital stay, reduced hospital costs, and increased patient satisfaction.

The ultrasound-guided erector spinae plane (ESP) block is a recent block described for various surgeries for postoperative analgesia. It is reported that it have an analgesic effect on somatic and visceral pain by affecting the ventral rami and rami communicantes that include sympathetic nerve fibres, as LA spreads through the paravertebral space. When performed bilaterally it has been reported to be as effective as thoracic epidural analgesia.

The transversus abdominis plane (TAP) block is a technique of locoregional anesthesia that blocks the sensorial afferent nerves localized between the transversus abdominis muscle and the internal oblique muscle.

In this study, the analgesic efficacy and duration of ultrasound (US) guided Erector spinea plane block and Transversus abdominis plane block when Lidocaine HCL is added as an adjuvant to bupivacaine will be compared.

DETAILED DESCRIPTION:
Sample size was calculated using Power Analysis and Sample Size software program (PASS) version 15.0.5 for windows (2017) using previous results with the mean opioid consumption in the first postoperative day as the primary outcome. Effect size of 0.5 (medium effect size) was calculated using the difference between the mean opioid consumption in TAB group (140 mg) and that in ESPB group (124.6 mg) with an estimated standard deviation of 30 in both groups. This study will add a control group in which only intravenous analgesics will be used; hence the aforementioned effect size was used for sample size calculation using a one-way ANOVA test. Sample sizes of 18 patients in each group are needed to achieve 90% power (1-β) to detect differences among the means using an F test with a 0.05 significance level (α). The size of the variation in the means is represented by the effect size f = σm / σ, which is 0.5. A 20% drop out is expected so the drop-out inflated sample size will be 23 patients in each group.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologist grade I-II

Exclusion Criteria:

* Patient refusal.
* Local skin infection and sepsis at the site of the block.
* Allergy to local anesthetic used.
* Hematological diseases
* Bleeding disease.
* Coagulation abnormality.
* Psychiatric disorders.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption | For 24 hours after performing block
  cumulative consumption of rescue opioids during the first postoperative day

SECONDARY OUTCOMES:
Duration of analgesia | for 24 hours after performing block
  the first time patient requests analgesia postoperatively
Postoperative visual analogue score | for 24 hours after performing block
  postoperative visual analogue score (VAS)which will be used to determine the postoperative pain levels in patients. ( 0 representing no pain and 10 is the worst imaginable pain) will be assessed at 2h, 4h,6h,12h,18h and 24h postoperative. Diclofenac75 mg IV and paracetamol 500 mg will be given to all patients in the three groups every 12 hours. If VAS is > 4 patient will receive pethidine 25 mg IV
Cortisol level | For one hour after performing block
  Cortisol level will be assayed in the serum
Heart rate | For 24 hours after surgery
  Changes in heart rate
Mean arterial blood pressure | For 24 hours after surgery
  Changes in mean arterial blood pressure
Peripheral oxygen saturation | For 24 hours after surgery
  Changes in peripheral oxygen saturation as measured with pulse oximetry
Nausea and vomiting | For 24 hour after surgery
  0: No nausea, 1: mild nausea, 2: moderate nausea, 3: severe nausea or vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa M Elbendary, MD, Study Chair — Anesthesia Department, Faculty of Medicine, Mansoura University
Locations (1):
- Hanaa M Elbendary, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Following completing recruiting and opening the dataset, the investigators would upload the raw data and results to the registry
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available following completing the study for life-long
Access Criteria: The data will be accessible to the investigators and PRS administrators with hiding the identifiers for the patients

REFERENCES:
- [Result] Mankikar MG, Sardesai SP, Ghodki PS. Ultrasound-guided transversus abdominis plane block for post-operative analgesia in patients undergoing caesarean section. Indian J Anaesth. 2016 Apr;60(4):253-7. doi: 10.4103/0019-5049.179451. PMID 27141108